CLINICAL TRIAL: NCT03075631
Title: Acute Pancreatitis Patient Registry To Examine Novel Therapies In Clinical Experiences 2
Acronym: APPRENTICE2
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Georgios Papachristou, Professor of Medicine, University of Pittsburgh
Other Study IDs: PRO15100089
Record Dates: First submitted 2017-02-02; First posted 2017-03-09 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens will be collected to look at biological measures.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with Acute Pancreatitis: Patients with Acute Pancreatitis
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaires

SUMMARY:
This study is an ancillary of APPRENTICE. This will be the international based study.

DETAILED DESCRIPTION:
This study is an ancillary of APPRENTICE. This will be the international based study. The initial study design with discussions about the different variables to be included into our prospective database started during 2014 PancreasFest held in Pittsburgh, PA in late July 2014 under the sponsorship of Collaborative Alliance for Pancreatic Education and Research (CAPER). Following this, a datasheet with variables was created, distributed through the initial participants, and further suggestions and edits were made. We now plan to move ahead with a web based seminar. All previous participants, as well as new investigators/centers that have shown interest in participating throughout the world will be invited.University of Pittsburgh will be responsible for collecting all required regulatory documents from other sites. Developing templates for questionnaires and other data collection forms. Will train approved sites on procedures. The coordinating center will be the recipient of de-identified data and will not be involved in the collection of data.

Note that copies of training records, licenses, certificates should be maintained in the study regulatory binder and are subject to audit by the Research Conduct and Compliance Office (RCCO).

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of AP based upon presence of two out of the three following criteria:

   1. Abdominal pain typical to AP
   2. Serum amylase or lipase levels more than three times the upper limit of normal
   3. Imaging findings suggestive of AP
2. Willingness to participate in the study and ability to sign informed consent by patient or his/her proxy (if unable to speak).

Exclusion Criteria:

1. Age under 18 years
2. Unwilling to provide consent by patient or his/her proxy
3. Presence of pancreatic cancer
4. Presence of chronic pancreatitis
5. Occurrence of AP following a multiple trauma episode
6. Having history of organ transplant
7. Presence of any cancer which required chemotherapy or radiation therapy in the past year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Acute Pancreatitis
Sampling Method: Probability Sample
Enrollment: 1183 (Actual)
Dates: Start 2015-12; Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with pancreatic necrosis as assessed by their clinical course. | 12 months
  Evaluation of the existing risks, predictive scores, and markers of severe disease.
Number of patients with persistent organ failure as assessed by their clinical course. | 12 months
  Evaluation of the current management and outcomes of acute pancreatitis around the world.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios I Papachristou, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Presbyterian, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
The results will be shared with the other IRB approved sites associated with this study.